CLINICAL TRIAL: NCT01261338
Title: Intervention to Reduce Body Burdens of PCBs in Residents of Anniston, Alabama
Acronym: PCBs
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10100801 1R21ES019206-01; 1R21ES019206-01 (NIH); 8 UL1 TR00007 (Other Grant/Funding Number: NCRR and NCATS)
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2016-12

CONDITIONS: Toxic Effect of Other Corrosive Organic Compounds
Keywords: PCBs; Olestra
MeSH Terms: interventions — sucrose polyester; Fat Substitutes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- olestra (Experimental): Non-absorbable fat administered in the form of 24 potato crisps per day (12 each with mid-day and evening meal) providing approximately 15g/day of olestra.
  Interventions: Drug: olestra
- Vegetable oil (Placebo Comparator): Absorbable fat administered in the form of 12 potato crisps per day (6 each with mid-day and evening meal) in order to match the caloric intake provided by the crisps with Olestra.
  Interventions: Drug: olestra

INTERVENTIONS:
Drug: olestra — non-absorbable dietary fat
  Other Names: Olean; non absorbable fat; fat substitute

SUMMARY:
Because of industrial pollution, a large number of people in Anniston, Alabama, have elevated body burdens of the class of compounds known as polychlorinated biphenyls (PCBs). There is evidence that these compounds are associated with risks to health including diabetes. There is also evidence that the consumption of a non-absorbable dietary fat can reduce the level of compounds like PCBs. This clinical trial will test the hypothesis that a non-absorbable dietary fat can reduce the levels of PCBs in subjects in Anniston.

DETAILED DESCRIPTION:
A clinical trial will be conducted which will test the use of a safe and minimally invasive dietary intervention to enhance the removal of toxic polychlorinated biphenyls (PCBs) from individuals with elevated levels of these compounds. To conduct this study, participants will be recruited and enrolled in Anniston, Alabama, a community in which a significant portion of the local population has been exposed to PCBs as a result of contaminated commercial waste. Many of the residents of Anniston currently have markedly elevated blood and adipose tissue PCB levels. In addition, these individuals have a several-fold increased prevalence of type-2 diabetes and are potentially at greater risk of other health disorders. .

A method was developed for adding a small amount of non-absorbable fat to the diet for use as a therapeutic tool which hastens the elimination of persistent lipophilic compounds, such as PCBs, in a safe manner. The rationale is based on the fact that once PCBs and other organochlorine pollutants enter the body, they circulate among several organs including the small intestine. Under normal circumstances, these compounds are reabsorbed from the intestine and returned to the blood, and are thus prevented from being excreted in the feces. The addition of a small amount of non-absorbable lipid in the diet provides a matrix for physically retaining the pollutants within the intestinal lumen, which then allows the pollutants to be excreted along with the lipid. Although the excretion on any given day is relatively small, the cumulative excretion over the course of a year becomes clinically significant. The Anniston population provides an ideal population to assess this intervention in a meaningful way, and we have allied with a local community group to assist in the recruitment of subjects and to carry out the relatively simple dietary manipulations required for this study.

A double-blind, placebo controlled study of a non-absorbable fat in subjects known to have elevated levels of PCBs will be conducted. The rate of change of the blood levels of PCBs in these subjects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Elevated blood level of PCBs

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weight-loss medication
* Gastrointestinal disease

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Jandacek, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- West Anniston Foundation, Anniston, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jandacek RJ, Heubi JE, Buckley DD, Khoury JC, Turner WE, Sjodin A, Olson JR, Shelton C, Helms K, Bailey TD, Carter S, Tso P, Pavuk M. Reduction of the body burden of PCBs and DDE by dietary intervention in a randomized trial. J Nutr Biochem. 2014 Apr;25(4):483-8. doi: 10.1016/j.jnutbio.2014.01.002. Epub 2014 Jan 29. PMID 24629911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-eight participants were recruited prior to April 2011.
Pre-assignment Details: Participants were randomized into groups of 14 each, to receive either olestra and vegetable oil.
Groups:
- Olestra: Non-absorbable fat
  olestra : non-absorbable dietary fat
- Vegetable Oil: absorbable fat
Period: Overall Study
Arm/Group | Olestra | Vegetable Oil
Started | 14 (One person in the olestra group started 4 months after the trial began.) | 14
Completed | 11 | 12
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olestra | Vegetable Oil | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.6) | 61.0 (5.7) | 60.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline for Total PCB Levels
Description: The outcome is the percent change in body burden of total PCB's measured over one year. Initially the percent of baseline is calculated as (value at one year / value at baseline) *100, then this is examined modeling over time as compared to the 100% at baseline.
Time Frame: one year
Population: Per protocol, based on elevated PCB levels
Measure: Mean (Standard Error); unit: % of baseline total PCBs
Arm/Group | Olestra | Vegetable Oil
Number analyzed (Participants) | 11 | 12
% of baseline total PCBs | 92 (3.4) | 96 (4.3)

2. Primary Outcome: Rate of Change of Lipid Adjusted PCB Levels
Description: This is a measure of the change in body burden of PCBs
Time Frame: One year
Population: All participants who completed the trial were analyzed.
Measure: Mean (Standard Error); unit: ng/g lipid/year
Arm/Group | Olestra | Vegetable Oil
Number analyzed (Participants) | 11 | 12
ng/g lipid/year | -0.0829 (0.0357) | -0.0413 (0.0408)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Olestra | Vegetable Oil
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/14
Other Adverse Events (participants affected / at risk) | 9/14 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olestra (N=14) | Vegetable Oil (N=14)
Hospitalized for heart catheter (Cardiac disorders) | 1 (1) | 0 (0) — Participant had a previous history of heart disease. There as no relationship to the study treatment.
Bleeding Ulcers (Gastrointestinal disorders) | 0 (0) | 1 (1) — Admitted to hospital
Chest pain and palpitations (Cardiac disorders) | 0 (0) | 1 (1) — Admitted to hospital
Heart stent replacement (Cardiac disorders) | 1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olestra (N=14) | Vegetable Oil (N=14)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (4)
Cold (General disorders) | 1 (1) | 0 (0)
Rash on body (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Irregular heartbeat (Cardiac disorders) | 0 (0) | 1 (1)
Pain in right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash on left and right anticubital area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection in lining of rib cage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Yeast Infection (Infections and infestations) | 1 (1) | 0 (0)
HGA1C elevated 6.4% (Endocrine disorders) | 1 (1) | 0 (0)
Cough (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No